CLINICAL TRIAL: NCT05567718
Title: The Relationship Between Fasting Time and Emergency Delirium in Pediatric Sedation Undergoing Magnetic Resonance Imaging
Brief Title: The Relationship Between Fasting Time and Delirium
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Neslihan Balkaya, medical doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2021/12/07
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Delirium; Sedation Complication; Magnetic Resonance Imaging; Fasting
Keywords: Emergence delirium; pediatric; preoperative fasting; magnetic resonance imaging
MeSH Terms: conditions — Delirium; Fasting; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Paediatric Anaesthesia Emergence Delirium scale — measure emergence delirium in children

SUMMARY:
We investigated the relationship between fasting times and delirium in children undergoing MRI under anesthesia. Paediatric Anaesthesia Emergence Delirium (PAED) scale, last oral intake time and type of food (solid-liquid) and fasting time, laryngospasm, desaturation (SpO2 <95%), bradycardia, allergy, nausea and vomiting were recorded.

ELIGIBILITY:
Inclusion Criteria:

* children between the age group 2-6 years of American Society of Anesthesiologists (ASA) physical status I or II
* Patients undergoing MRI under sedation

Exclusion Criteria:

* ASA 3-4-5
* under 2 years old, over 6 years old
* cognitive or psychological disorder
* serious central nervous system diseases, including a brain tumor or uncontrolled seizures
* type 1 diabetes
* detection of ≤ 50 mg/dl in fasting blood glucose measurement
* whose parents did not want to participate in the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children between the age group 2-6 years of American Society of Anesthesiologists (ASA) physical status I or II, patients undergoing MRI under sedation
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium scale | during the procedure
  to measure delirium using the scale

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek Ihtisas Training and Research Hospital, Yıldırım, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No